CLINICAL TRIAL: NCT05274672
Title: Does Post-operative Antibiotic Prophylaxis Reduce Urinary Tract Infection Rates After Holmium Laser Enucleation of Prostate? a Prospective Randomized Multi-center Study
Brief Title: Role of Prophylactic Postoperative Antibiotics in HoLEP
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment.
Sponsor: Baylor Research Institute (Other)
Collaborators: Albert Einstein Healthcare Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 022-046
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Benign Prostatic Hyperplasia; Urinary Tract Infections
Keywords: HoLEP; Prophylactic antibiotics; Urinary tract infection
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Tract Infections | interventions — Nitrofurantoin; Cephalexin; Trimethoprim, Sulfamethoxazole Drug Combination; Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: Study to be multi-institutional, double armed, randomized controlled trial between Baylor Scott and White medical center in Temple, Texas and Albert Einstein Medical Center in Philadelphia.
  The study will include 100 patients who will have HoLEP in the 2 centers within almost one year, between March 2022 and March 2023. Patients will be randomized in to 2 groups:
  * Group I: Experimental Group (not receiving antibiotics).
  * Group II: Control Group (receiving 3 days of antibiotics after surgery)
  Each center will have a study coordinator (resident and/or fellow) that will be responsible for randomization using closed envelope technique.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients not receiving postoperative antibiotics (Experimental): Patients who will not receive prophylactic postoperative antibiotics after HoLEP.
  Interventions: Procedure: Holmium Laser Enucleation of prostate
- Patients receiving postoperative antibiotics (Active Comparator): Patients who will receive3 days prophylactic postoperative antibiotics after HoLEP.
  Interventions: Drug: Nitrofurantoin; Drug: Cephalexin; Drug: Sulfamethoxazole Trimethoprim Combination; Drug: Ciprofloxacin; Procedure: Holmium Laser Enucleation of prostate

INTERVENTIONS:
Drug: Nitrofurantoin — Prophylactic postoperative antibiotic use
  Other Names: Macrobid
  Arms: Patients receiving postoperative antibiotics
Drug: Cephalexin — Prophylactic postoperative antibiotic use
  Other Names: Keflex
  Arms: Patients receiving postoperative antibiotics
Drug: Sulfamethoxazole Trimethoprim Combination — Prophylactic postoperative antibiotic use
  Other Names: BACTRIM
  Arms: Patients receiving postoperative antibiotics
Drug: Ciprofloxacin — Prophylactic postoperative antibiotic use
  Other Names: Cipro
  Arms: Patients receiving postoperative antibiotics
Procedure: Holmium Laser Enucleation of prostate — Endoscopic transurethral Holmium Laser enucleation of enlarged prostate followed by morcellation of prostatic tissue
  Other Names: HoLEP

SUMMARY:
The purpose of this study is to investigate whether prescribing a 3-day course of antibiotics after Holmium laser enucleation of the prostate (HoLEP) reduces the risk of urinary tract infection. The findings of this trial will have a major impact on clinical practice to either justify the prescription of antibiotics after HoLEP or give urologists more confidence in not prescribing antibiotics prophylactically after HoLEP.

DETAILED DESCRIPTION:
Systemic antibiotic usage is the primary driver of antimicrobial resistance both in the index patient and the community. Limiting antibiotic use to indicated patients helps reduction of the risks of antimicrobial overuse, which include associated adverse events, development of multidrug resistant (MDR) organism strains, and increased health-related community burden. (1-3) Holmium laser enucleation of the prostate (HoLEP) has been increasingly used as an effective minimally invasive procedure for the management of enlarged prostate. (4) Most guidelines currently recommend the use of single-dose antibiotic prophylaxis prior to all transurethral procedures for the treatment of benign prostatic hyperplasia including HoLEP. (2,3) Although, most surgeons who perform HoLEP usually extend the antibiotics prophylaxis to 3-7 days or more after HoLEP to avoid the incidence of urinary tract infection. Currently no literature that supports the benefit of prescribing antibiotics routinely to all patients after HoLEP. (5, 6) 2. Significance: This clinical trial will provide insight into the benefit of prescribing antibiotics after HoLEP. This study can be practice-changing for urologists who perform HoLEP as it will decrease the prescription of unnecessary antibiotics. This has major implications for antibiotic stewardship in the field of urology.

3. Objectives & Specific Aims: The purpose of this study is to investigate whether prescribing a 3-day course of antibiotics after HoLEP reduces the risk of urinary tract infection. The findings of this trial will have a major impact on clinical practice to either justify the prescription of antibiotics after HoLEP or give urologists more confidence in not prescribing antibiotics prophylactically after HoLEP.

The specific aims of this study are:

1. Avoid the possible unnecessary generalized prolonged antibiotic prophylaxis in patients with HoLEP.
2. Identify the patient and procedure factors that increase the incidence of postoperative urinary tract infection.
3. Possible selection of patients who can benefit from prolonged antibiotic prophylaxis.
4. Help changing the urology practice towards more antibiotic stewardship.

4. Methodology: 4.1 Study Design.

Study to be multi-institutional, double armed, randomized controlled trial at Baylor Scott and White medical center in Temple, Texas and Albert Einstein Medical Center in Philadelphia.

The study will include 100 patients who will have HoLEP in the two centers within almost one year, between March 2022 and March 2023.

All patients will receive a single perioperative antibiotics per the American urological association guidelines. Patients will be randomized in to 2 groups:

* Group I: Experimental Group (not receiving antibiotics).
* Group II: Control Group (receiving three days of antibiotics after surgery)

Each center will have a study coordinator (resident and/or fellow) that will be responsible for randomization using the closed envelope technique.

4.2 Procedures/Methods.

Each patient's chart in the study will be subjected to analysis of:

1. Preoperative assessment:

   * Detailed history and physical examination.
   * Investigations:

     * Routine laboratory investigations, urine analysis and culture, serum PSA.
     * IPSS, Q-max, and PVR
2. Operative details:

   * Operative time, prostate volume
   * Estimated blood loss
   * Any intraoperative complications.
3. Postoperative assessment:

During early postoperative follow up, the patient will be assessed for:

* Irritative voiding symptoms, urinary urgency, urinary frequency, and urinary incontinence.
* IPSS, Quality of life (QOL)
* Assessment of PVR.

ELIGIBILITY:
Inclusion Criteria:

* Men > 40 years old with moderate to severe lower urinary tract symptoms due to benign prostatic hyperplasia (BPH).
* Patient with negative preoperative urine culture.

Exclusion Criteria:

* Patients with history of recurrent urinary tract infection or uro-sepsis.
* Patient with preoperative infections
* Patient with indwelling urethral catheter
* Patient doing continuous intermitted catheterization (CIC)

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The Benign prostatic pathology is applicable only in male patients.
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
the rates of urinary tract infection within the 30-day post-operative period after HoLEP | within 30 days after HoLEP
  A urinary tract infection is defined as a positive urine culture .

SECONDARY OUTCOMES:
The incidence of irritative voiding symptoms after HoLEP and all the other urinary functional outcomes. | 6 months
  Irritative voiding symptoms, postoperative hematuria, incontinence, urethral stricture, need for re-catheterization.

CONTACTS AND LOCATIONS:
Overall Officials: Marawan M. El Tayeb, MD, Principal Investigator — Baylor Scott and White Health Medical Center
Locations (2):
- United States (2):
  - Einstein Healthcare network, Philadelphia, Pennsylvania
  - Baylor Scott and White, Temple, Texas

IPD SHARING:
Plan to Share IPD: No
All the published material will keep human information in an unidentifiable manner.

REFERENCES:
- [Background] Tennyson LE, Averch TD. An Update on Fluoroquinolones: The Emergence of a Multisystem Toxicity Syndrome. Urol Pract. 2017 Sep;4(5):383-387. doi: 10.1016/j.urpr.2016.08.004. Epub 2016 Oct 24. PMID 37592645
- [Background] Lightner DJ, Wymer K, Sanchez J, Kavoussi L. Best Practice Statement on Urologic Procedures and Antimicrobial Prophylaxis. J Urol. 2020 Feb;203(2):351-356. doi: 10.1097/JU.0000000000000509. Epub 2019 Aug 23. PMID 31441676
- [Background] Ivan SJ, Sindhwani P. Comparison of guideline recommendations for antimicrobial prophylaxis in urologic procedures: variability, lack of consensus, and contradictions. Int Urol Nephrol. 2018 Nov;50(11):1923-1937. doi: 10.1007/s11255-018-1971-1. Epub 2018 Aug 25. PMID 30145652
- [Background] Das AK, Teplitsky S, Humphreys MR. Holmium laser enucleation of the prostate (HoLEP): a review and update. Can J Urol. 2019 Aug;26(4 Suppl 1):13-19. PMID 31481144
- [Background] Ishikawa K, Maruyama T, Kusaka M, Shiroki R, Hoshinaga K. [The state of antimicrobial prophylaxis for holmium laser enucleation of the prostate : HoLEP and the results of a questionnaire survey]. Hinyokika Kiyo. 2011 Oct;57(10):539-43. Japanese. PMID 22089150
- [Background] Davuluri M, Bernstein AP, Fram E, Watts KL. Variations in Perioperative Antibiotic Prescriptions Among Academic Urologists After Ambulatory Endoscopic Urologic Surgery: Impact on Infection Rates and Validation of 2019 Best Practice Statement. Urology. 2020 Dec;146:101-106. doi: 10.1016/j.urology.2020.07.049. Epub 2020 Aug 8. PMID 32777364